CLINICAL TRIAL: NCT06898138
Title: Acute Stimulation for the Modulation of Epileptic Events with a Closed-Loop Brain Interchange System in Drug Resistant Epilepsy
Brief Title: Acute Stimulation and Modulation of Stereotyped High-Frequency Oscillations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Baylor College of Medicine (Other); CorTec GmbH (Unknown)
Responsible Party: Principal Investigator, Nuri F. Ince, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-012951; UH3NS117944 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: neuromodulation; HFO; Epilepsy; Machine Learning; Closed-Loop
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: In a multi-phase structure, the project will investigate the feasibility of recording the HFOs with the BIC system (Cortec, Germany) and then delivering closed-loop stimulation.
  In this phase of the project, the feasibility of delivering of closed-loop stimulation with the implantable system will be tested. For this 8 subjects will be recruited.
  Therefore, in this phase of the study, a total 8 subjects will be recruited in a sequential fashion to test device feasibility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Epilepsy (Experimental): Patients with drug resistant epilepsy undergoing a surgical evaluation in the epilepsy monitoring unit
  Interventions: Device: Brain Interchange System

INTERVENTIONS:
Device: Brain Interchange System — The CorTec Brain Interchange (BIC) is an implantable system with sensing and stimulation capability dedicated to promoting brain computer interface and closed-loop neuromodulation research. It is an externally powered implant which can provide neural data to a nearby computing station (communication unit connected to a personal computer) continuously. In return, computing station controls the implant e.g. for generating therapeutic electrical stimulation to the brain. It is expected that BIC will catalyze translational applications of electroceuticals in human subject by making the neural data immediately available as well as permit the investigation of novel closed-loop neuromodulation applications.

SUMMARY:
Overall, this study will investigate the functional utility of stereotyped HFOs by capturing them with a new implantable system (Brain Interchange - BIC of CorTec), which can sample neural data at higher rates >=1kHz and deliver targeted electrical stimulation to achieve seizure control. In contrast to current closed-loop systems (RNS), which wait for the seizure to start before delivering stimulation, the BIC system will monitor the spatial topography and rate of stereotyped HFOs and deliver targeted stimulation to these HFO generating areas to prevent seizures from occurring. If the outcomes of our research in an acute setting become successful, the investigators will execute a clinical trial and run the developed methods with the implantable BIC system in a chronic ambulatory setting.

DETAILED DESCRIPTION:
High-frequency oscillations (HFOs) of intracranial EEG (iEEG) have the potential to identify the surgical resection area/seizure onset zone (SOZ) in patients with drug-resistant epilepsy. However, multiple reports indicate that HFOs can be generated not only by epileptic cerebral tissue but also by non-epileptic sites often including eloquent regions such as motor, visual, and language cortices. In this project, the initial evidence of a recurrent waveform pattern is presented that may be sufficient to distinguish pathological HFOs from physiological ones. Specifically, the investigators show that the SOZ repeatedly generates sets of stereotypical HFOs with similar waveform morphology whereas the events recorded from out of SOZ were irregular. This morphological pattern served as a robust neurobiomarker to isolate SOZ from other brain areas in multiple patients consistently. While these promising preliminary results are in place, the functional utility of stereotyped HFOs in a closed-loop seizure control system remains unknown. As of today, not much is known whether the stereotyped HFOs generated by the SOZ can be detected with an implantable system. If this can be achieved, then HFOs can be strategically translated as a neurobiomarker into closed-loop seizure control applications. The investigators hypothesize that pathologic stereotyped HFOs can be captured with the implantable Brain Interchange (BIC) system of CorTec and spatial topography of these events can be utilized by the implantable system to deliver targeted electrical stimulation to achieve seizure control. Using an acute setup within the epilepsy monitoring unit (EMU), this project will investigate the feasibility of capturing stereotyped HFO events using the new BIC system and compare the detection results to those obtained with the commercially available amplifier (Aim-1). If the first phase (Aim-1) of the study becomes successful, later in the second phase (Aim-2), once again in the EMU, the investigators will deliver targeted electrical stimulation to those brain sites associated with stereotyped HFOs using the BIC.

During the entire study, the BIC system will not be implanted but used externally to assess the neural data through externalized electrodes and then deliver closed-loop stimulation. If the outcomes of the research in an acute setting become successful, the investigators will execute a clinical trial and run our methods with the implanted BIC system in a chronic ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medically refractory epilepsy, who have been deemed appropriate candidates for intracranial EEG monitoring
* Adult men and women (18≤ age <70 years)
* Children (3≤ age <18 years)
* Includes women and minorities

Exclusion Criteria:

• Subjects will be excluded if their condition makes them unable to continue with recordings.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Detection of Stereotyped HFOs | Within the first 3 years of the project
  Outcome-2 will test the feasibility of capturing stereotyped HFO (sHFO) with the BIC system in the EMU setting. Once the feasibility of robust data transmission as listed in (Outcome-1) is tested, the neural activity will be recorded over 24 hours using the BIC system from 10 patients. The hardware will not be implanted but used externally to record the neural data. Then, the research team will compare whether the sHFO detection and SOZ localization accuracy is significantly different between the BIC and FDA approved amplifier. If the investigators can detect stereotyped HFOs with a rate not less than 75% of FDA approved clinical amplifier and predict the SOZ in 8/10 patients, then the research team will move to the second phase of the project to test Outcome-3. Outcome-2 tests the feasibility of capturing relevant neural events with the external BIC system and compares the recording quality to the FDA approved amplifiers. Outcome-2 does not test any health-related outcome.
Feasibility of Delivering Closed-Loop Stimulation | In the 4th and 5th years of the project
  Outcome-3 will test the feasibility of delivering of closed-loop stimulation with the BIC system. If the detection of sHFO with the BIC system is feasible (Outcome-2), the investigators will start to test the online methods on the previously recorded datasets to isolate sHFOs in streaming iEEG/ECoG. Using the computer in the loop real-time system and the BIC, in the last 2 years, closed-loop stimulation will be delivered. In total 8 patients will be recruited for this particular purpose. Targeted stimulation will be delivered to those channels associated with sHFOs and other areas which are not associated with sHFOs. The research team will test if the device can deliver stimulation to selected channels without any failure. The BIC system will not be implanted but used externally to deliver the stimulation. Outcome-3 does not test whether the system can control the seizures of the patients. It only investigates the feasibility of delivering closed-loop stimulation.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Intracranial EEG + ECoG recorded from patients with epilepsy will be shared. The electrical signs of neural activity will be collected in the EMU for 24hrs. One stream of data will be digitized at 1kHz with 16bit resolution with the BIC system and the other stream with least a 2 kHz sampling frequency to capture HFOs reaching up to 500Hz.
  Additionally, the closed-loop stimulation data with stimulation parameters including onset, duration, frequency, pulse width, and amplitude information will be shared. All collected data will be de-identified prior to data exchange. Patient data will be provided in a coded format that protects patient identities but will contain diagnosis (signs/symptoms), interventions including technical observations, diagnostic tests/results, and patient outcomes.
  Information about the device delivering therapy including device serial numbers, device model numbers, date of the event, and country/state of the event will be annotated with the data and therapy
Time Frame: Every 6 months
Access Criteria: Data Archive for the BRAIN Initiative (DABI) - invasive human neurophysiology (including EEG, ECoG, LFP, single unit)
URL: http://dandiarchive.org

REFERENCES:
- [Background] Ayyoubi AH, Fazli Besheli B, Quach MM, Gavvala JR, Goldman AM, Swamy CP, Bartoli E, Curry DJ, Sheth SA, Francis DJ, Ince NF. Benchmarking signal quality and spatiotemporal distribution of interictal spikes in prolonged human iEEG recordings using CorTec wireless brain interchange. Sci Rep. 2024 Feb 8;14(1):2652. doi: 10.1038/s41598-024-52487-5. PMID 38332136